CLINICAL TRIAL: NCT02141126
Title: Can Lower Limb Resistance Training Improve Strength, Muscle Mass and Functional Outcomes in Older Inpatients in a Post-acute Rehabilitation Unit? A Randomised Controlled Feasibility Study
Brief Title: Lower Limb Resistance Training in Older Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: St. James's Hospital, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCSI-SJH; RCSI-SJH-MISA (Other: RCSI-SJH-MISA); RCSI-SJH-MISA-2013 (Other: RCSI-SJH-MISA-2013)
Record Dates: First submitted 2014-01-06; First posted 2014-05-19 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2017-04

CONDITIONS: Muscle Weakness
Keywords: Older adults; Strength training; Muscle mass; Function; Inpatients
MeSH Terms: conditions — Muscle Weakness | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Feasibility study Randomised and controlled
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance training (Experimental): Usual care and resistance exercises.
  Interventions: Other: Resistance training
- Usual care (Other): Usual inpatient physiotherapy
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Resistance training — Usual physiotherapy care and twice weekly tailored and progressive resistance lower limb exercises Circuit-type format, sessions will last 35 minutes and will include a warm-up and cool-down period. Exercises tailored to each patient and will use ankle weights as the resistance, using 65-75% of their 1-Repetition Maximum. Intervention will last for 6 weeks.
  Arms: Resistance training
Other: Usual care — Standard inpatient 'usual care' physiotherapy
  Arms: Usual care

SUMMARY:
The primary aim of this feasibility study is to evaluate the feasibility of delivering a PRT programme in an inpatient older person rehabilitation setting and to describe changes in lower limb strength and physical function following six weeks of resistance training and routine physiotherapy versus a control group of routine physiotherapy only in an older inpatient population.

DETAILED DESCRIPTION:
This is a prospective, single blinded, randomised controlled feasibility study recruiting consecutive appropriate patients in this post-acute rehabilitation unit.

Feasibility outcomes including safety, recruitment, measurements, adherence, retention and satisfaction will be evaluated. There are two groups (i) exercise intervention and (ii) control. It will not be possible to blind the treating physiotherapist or the patient to the exercise intervention; hence the single (assessor) blinded design.

The study will be based in St James's Hospital, Dublin. Assessments and the delivery of the exercise intervention will be conducted in the Physiotherapy department.

Patients will be recruited in the inpatient setting. Appropriate patients will be approached, and the intervention explained to them. The patient will be given an information leaflet and 24-hours to consider involvement in the study

ELIGIBILITY:
Inclusion Criteria:

* Patients, male and female elderly inpatients 65 years.
* Patients must be medically stable.
* Patients who are able to follow one-stage commands.
* Patients must be able to give informed consent.

Exclusion Criteria:

* Unstable medical condition.
* Patients who are unable to follow one-stage commands.
* Acute pain or fracture
* Patients who are unable to stand or require more than assistance of two staff to mobilise/transfer.
* Patients who have been admitted with a recent diagnosis of stroke, due to their varying patterns of recovery.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Lower limb dynamometry | Baseline, Week 6
  Lower limb dynamometry will be measured using the Power Track II Commander by J-Tech Medical. A previous study in this rehabilitation unit has determined that this is a reliable measure of lower limb strength in this population. The primary outcome measurement will be quadriceps muscle strength.

SECONDARY OUTCOMES:
Functional mobility using the Timed Up and Go (TUG) | Baseline, Week 6
  Functional mobility using the Timed Up and Go (TUG) - this is a test of basic functional mobility for frail elderly people. The patient is asked to stand up from a chair, walk three metres, turn around and return to the chair, while being timed by the assessor.
Six Minute Walk Test (6MWT) | Baseline, Week 6
  Six Minute Walk Test (6MWT) - this is a performance-based test. The distance walked in six minutes is measured and reported in metres or feet and is an indication of exercise tolerance.
EuroQol-5D (EQ-5D) | Baseline, Week 6
  EuroQol-5D (EQ-5D) - measures health related quality of life, it contains a visual analogue scale (0 to 100, representing dead to excellent health state) and five items: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Canadian Study of Health and Ageing Clinical Frailty Scale (CFS) | Baseline, Week 6
  Canadian Study of Health and Ageing Clinical Frailty Scale (CFS) - this is a measure of frailty based on clinical judgement. It is an ordinal scale which ranges from 1 to 7. Reliability and validity have been proven in an older population (Rockwood et al, 2005).

OTHER OUTCOMES:
Height and Weight and BMI | Baseline, Week 6
  Height will be measured from ulna length (BAPEN, 2004), weight will be measured using body composition scales, and body mass index (BMI) calculated using these measures.
Skeletal muscle mass | Baseline, Week 6
  Skeletal muscle mass will be calculated using a validated equation based on measured bioimpedance from the body composition scales (Janssen J Appl Phil 2000).
Grip Strength | Baseline, Week 6
  Grip strength will be measured using a handgrip dynamometer on the non-dominant arm (Clinifeed/Roussel dynamometer).

CONTACTS AND LOCATIONS:
Overall Officials: Sinead Coleman, MSc, Principal Investigator — St James's Hospital, James's Street, Dublin 8, Ireland; Frances Horgan, PhD, Principal Investigator — Royal College of Surgeons in Ireland; Niamh Murphy, MSc, Study Director — St James's Hospital, James's Street, Dublin 8, Ireland; Gareth Clifford, MSc, Study Director — St James's Hospital, James's Street, Dublin 8, Ireland; David Robinson, MD, Study Director — St James's Hospital, James's Street, Dublin 8, Ireland; Conal Cunningham, MD, Study Director — St James's Hospital, James's Street, Dublin 8, Ireland
Locations (1):
- Physiotherapy Department, St James's Hospital, James's Street, Dublin 8, Ireland, Dublin, Ireland